CLINICAL TRIAL: NCT05380310
Title: Impact on the Time to Diagnosis of Serious Post-operative Complications of Continuous, Individualised, Alert Monitoring of SpO2, Heart Rate and Respiratory Rate by a Controlled Connected Medical Device (SMART ANGEL Intra )
Brief Title: Impact on the Time to Diagnosis of Serious Postoperative Complications by a Controlled Connected Medical Device
Acronym: SMARTANGEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Evolucare Technologies (Industry); InES - Innovation Electronic Software (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: APHP210932; N° IDRCB (Other: 2021-A01759-32)
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Medical Device
Keywords: Connected Medical Device; Time to diagnosis; Post-operative mortality; "SMART ANGEL intra-hospital" system

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active alerts (Experimental): "SMART ANGEL Intra-hospital" System with active alerts
  Interventions: Device: Active "SMART ANGEL" solution
- Inactive alerts (Active Comparator): "SMART ANGEL Intra-hospital" System with inactive alerts
  Interventions: Device: Inactive "SMART ANGEL" solution

INTERVENTIONS:
Device: Active "SMART ANGEL" solution — Nurse intervention according to the alert level + traditional monitoring
  Arms: Active alerts
Device: Inactive "SMART ANGEL" solution — No alert + traditional monitoring + alert in case of imminent life threat
  Arms: Inactive alerts

SUMMARY:
Post-operative mortality in case of scheduled surgery is 3% in France (Lancet 2013) mainly due to cardiovascular or respiratory complications, by decompensation of pre-existing pathologies.

Complications due to the medical practice are the third cause of morbidity (BMJ, 2016). More than half are preventable and are mainly observed in surgical patients. In conventional hospitalization, excluding intensive care, monitoring is done discontinuously for most of the patients, which does not allow early diagnosis of a vital cardiovascular or respiratory failure.

Diagnosis and late treatment do not allow good recovery. The early identification of a vital failure by the continuous monitoring of three simple physiological parameters (SpO2, heart rate and respiratory rate) would allow faster management by the hospital staff and a reduction in immediate and possibly delayed postoperative mortality.

DETAILED DESCRIPTION:
The challenge of this research is to transpose in an ordinary hospitalization unit the continuous monitoring of vital functions carried out in intensive care by the continuous measurement of simple parameters using the "SMART ANGEL Intra-hospital" System's (connected medical devices and alerts).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients receiving a scheduled non-ambulatory surgical or interventional procedure
* Affiliation to a social security scheme, beneficiary or entitled person (excluding AME)
* Patient's written consent or of the trusted person in case of physical incapacity

Exclusion Criteria:

* Inclusion in emergency situations
* ASA1 patient (without associated pathology)
* Patient with a multi-drug resistant germ in isolation
* Known linguistic inability of the patient to understand the study
* Known pregnancy or breastfeeding woman
* Patients with implantable pacemakers, implantable defibrillators or neurostimulators.
* Person under legal protection or unable to give consent
* Person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Difference in response times for nurses | between inclusion visit and day 30
  Difference in response times between the two groups as measured by the difference between the exact time of occurrence of the complication and the time of caregiver intervention.

SECONDARY OUTCOMES:
Mortality during hospitalisation | between inclusion visit and day 30
  Within 30 days of the intervention
Mortality within 30 days of surgery | between inclusion visit and day 30
Percentage of transfers to intensive care unit | between inclusion visit and day 30
Length of stay | between inclusion visit and day 30
ICU length of stay | between inclusion visit and day 30
Rate of calls to the doctor on duty | between inclusion visit and day 30
Percentage of re-hospitalization within 30 days | between inclusion visit and day 30
Percentage of hospitalisations in follow-up care and rehabilitation care units | between inclusion visit and day 30
Percentage of patients managed at home | between inclusion visit and day 30
False positive rate | between inclusion visit and day 30
  Alert without complication for the patient
Incremental cost-effectiveness ratio | between inclusion visit and day 30
Patient acceptability | between inclusion visit and day 30
  Quantitative and qualitative assessment of the device's usability by the patient via Questionnaire and interview
Acceptability of care teams | between inclusion visit and day 30
  Questionnaire and interview

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MARTY, MD,PHD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France